CLINICAL TRIAL: NCT01374893
Title: Effects of an Intrahospital Exercise Program in Functional Capacity of Old Inpatients
Brief Title: Physical Training in Hospitalized Elderly
Acronym: AGECAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Jose Antonio SERRA-REXACH (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Jose Antonio SERRA-REXACH, MD PhD, head of the Geriatrics Department, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HGUGregorioMaranon
Record Dates: First submitted 2011-06-09; First posted 2011-06-16 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Functional Impairment
Keywords: Function, hospitalization, elderly
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Active Comparator)
  Interventions: Behavioral: Exercise
- Control group (Placebo Comparator): Usual care
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Exercise — The intervention group will perform the multi-session per day training program
  Arms: Exercise
Behavioral: Control — Usual care
  Arms: Control group

SUMMARY:
Background The Activity in GEriatric acute CARe (AGECAR) is a randomized control trial to assess the effectiveness of an intrahospital strength and walk program during short hospital stays for improving functional capacity of patients aged 75 years or older.

DETAILED DESCRIPTION:
Objective: The main objective of this study is to assess whether an inpatient exercise program, beyond other components of interdisciplinary care, could reduce hospital associated disability (HAD) in medical patients aged 75 years and older admitted to an acute care for elders (ACE) unit.

Population: The reference population will be patients aged 75 years and older admitted to the ACE unit from the emergency department. This study will include only patients discharged alive. Exclusion criteria include patients fully dependent at baseline, unable to sign informed consent, unstable medical condition, short stay (<3 days), end stage illness.

Interventions: Patients will be randomly assigned to a control or an intervention group. Participants allocated to the control group will receive usual care in the ACE unit with actions directed to prevent delirium and functional decline. The intervention group, in addition to the usual care, will receive an exercise program. Briefly, this program consisted of strengthening of lower limbs muscles, and walking, daily from Monday to Friday.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include approximately 150 elderly people aged 75 years or older recruited from patients admitted into the Geriatrics Department of the Hospital General Universitario Gregorio Marañón (Madrid, Spain).
* Able to ambulate, with or without personal/technical assistance.
* Able to communicate.
* Informed consent: Must be capable and willing to provide consent.

Exclusion Criteria:

* Duration of hospitalization < 72 hours
* Any factor precluding performance of the physical training program or testing procedures as determined by the attending physician. These factors include, but are not limited to the following:
* Terminal illness.
* Myocardial infarction in the past 3 months.
* Not capable of ambulation.
* Unstable cardiovascular disease or other medical condition.
* Upper or lower extremity fracture in the past 3 months.
* Severe dementia.
* Unwillingness to either complete the study requirements or to be randomised into control or intervention group.
* Presence of neuromuscular disease or drugs affecting neuromuscular function.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 260 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2014-10-01 (Actual); Study Completion 2014-10-01 (Actual)

PRIMARY OUTCOMES:
Recover basal functional capacity | During hospital stay, from admission (first evaluation) until hospital discharge (second evaluation, and 3-months postdischarge (last evaluation).
  Changes in the number of Activities of daily living (ADLs) that the patients could perform independently. The six basic ADLs include: bathing, dressing, toileting, transferring, continence, and eating. For each ADL, a score of 0 is assigned for dependence and 1 for independence. A summary scale is constructed by summing the individual ADLs (range of 0-6). Recovery is defined as performance that is at least as good at discharge or 3-months postdischarge as it was at baseline.

SECONDARY OUTCOMES:
Ability to walk independently | During hospital stay, from admission (first evaluation) until hospital discharge (second evaluation, and 3-months postdischarge (last evaluation).
  Changes in Functional Ambulation Classification (FAC) scale as one of five functional levels of ambulation (range of 0-4). A score of 0 is assigned if the patient cannot walk, one if the patient requires continuous manual contact to support the body, 2 for light or intermittent manual contact to assist balance, 3 for independent but supervised ambulation, and 4 for independent ambulation on level surfaces or stairs. Recovery is defined as performance that is at least as good at discharge or 3-months postdischarge as it was at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Serra, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (1):
- Geriatric Department, Hospital General Universitario Gregorio Marañón, Madrid, Spain

REFERENCES:
- [Derived] Ortiz-Alonso J, Bustamante-Ara N, Valenzuela PL, Vidan-Astiz M, Rodriguez-Romo G, Mayordomo-Cava J, Javier-Gonzalez M, Hidalgo-Gamarra M, Lopez-Tatis M, Valades-Malagon MI, Santos-Lozano A, Lucia A, Serra-Rexach JA. Effect of a Simple Exercise Program on Hospitalization-Associated Disability in Older Patients: A Randomized Controlled Trial. J Am Med Dir Assoc. 2020 Apr;21(4):531-537.e1. doi: 10.1016/j.jamda.2019.11.027. Epub 2020 Jan 20. PMID 31974063
- [Derived] Fleck SJ, Bustamante-Ara N, Ortiz J, Vidan MT, Lucia A, Serra-Rexach JA. Activity in GEriatric acute CARe (AGECAR): rationale, design and methods. BMC Geriatr. 2012 Jun 9;12:28. doi: 10.1186/1471-2318-12-28. PMID 22682063